CLINICAL TRIAL: NCT03716154
Title: Clinical Effectiveness of Diode Laser as an Adjunct in the Treatment of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JUSTShbool1
Record Dates: First submitted 2018-10-08; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: split mouth
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRP and diode laser (Experimental): In a split mouth design either left or right sites randomly treated by SRP and diode laser as an adjunct
  Interventions: Radiation: Diode laser
- SRP alone (No Intervention): The other sites in the other side will be treated by SRP alone

INTERVENTIONS:
Radiation: Diode laser — Diode laser 810nm, 2W, 20sec, 20 HZ
  Arms: SRP and diode laser

SUMMARY:
a randomized controlled single-blinded study. the hypothesis of this clinical trial is that disjunctive use of diode laser improve the clinical parameters of periodontists , and there are significant difference between the conventional treatment and diode laser as an adjunct

DETAILED DESCRIPTION:
A total of 240 sites with deep pocket in 30 systemically healthy patients with chronic periodontitis, from subjects attending Jordan University of Science and Technology (JUST) Postgraduate Dental Clinic (PDC), the age range were (28-55) year, between Apr 2017 and Oct 2017. Those patients were enrolled in a randomized controlled single-blinded study. For each patient, full medical and dental history and periodontal examination were recorded. Clinical parameters such as pocket depth (PD), clinical attachment loss (CAL), gingival index (GI) and plaque index (PI) were evaluated at the baseline. All Patients underwent initial periodontal therapy; SRP which was performed using a sonic device and hand instruments and the sites were divided randomly into two groups SRP alone and SRP with adjunctive diode 810 nm laser in the contralateral sites in the same jaw. The Clinical parameters have been re-evaluated at 1, 3 and 6 months to test the effectiveness of (810 nm, 2 W, pulsed mode, for 20 sec) in treatment of CP. Diode laser therapy was applied to periodontal pockets in the same day of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients having periodontitis in at least two quadrants each quadrant should have at least 4 sites with PD >4mm.
* Both male and female patients.
* Patient who are ready to cooperate with diode laser treatment.
* Patient who can comply with 3 visits for follow up (three times).

Exclusion Criteria:

* Subjects with systemic diseases that may interfere with wound healing (such as diabetes) or any systemic disease that complicates the treatment.
* Pregnant women and breast feeding.
* Smokers, alcohol or drug dependent.
* Patients who received any form of periodontal treatment within the last 6 months.
* Patients who are currently taking or were on antibiotic treatment within the last 6 months.
* Presence of faulty restoration at teeth involved in the disease.
* Teeth indicated for extraction at sites that will be part of the study.
* Patient under 18 years of age.

Ages: 28 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Probing depth (PD) in millimeter (mm), clinical attachment loss (CAL) in millimeter (mm) | Change from baseline to 1 month in PD and CAL, change from baseline to 3 month in PD and CAL ,change from baseline to 6 month in PD and CAL
  PD its the distance from gingival margin to the base of the pocket in millimeter (mm) CAL the recession is added to the PD in millimeter (mm)

OTHER OUTCOMES:
GI index score ,PI index score | Change from baseline in GI and PI at 1 month, change from baseline in GI and PI at 3 month, Change from baseline in GI and PI at 6 month
  GI index score:
  0 = normal gingiva (pink, scalloped margin, pin pointed papilla, thin buccal and lingual margin);
  1. = mild inflammation (slight changes in color, slight edema, no bleeding on probing);
  2. = moderate inflammation (redness, edema, bleeding on probing)
  3. = severe inflammation (marked redness, edema, ulceration, spontaneous bleeding).
  PI index score:
  0 = no plaque in the gingival area
  1. = a film of plaque adhering to the gingival margin and adjacent area of the tooth. The plaque may be only recognized by running a probe across the tooth surface.
  2. = moderate accumulation of soft debris within the gingival pocket on the gingival and/or on the tooth surface, which can be seen by naked eye.
  3. = abundance of soft matter within the gingival pocket and /or on the gingival margin and adjacent tooth surface.

CONTACTS AND LOCATIONS:
Overall Officials: rola A alhabashneh, prof, Study Director — Jordan University of Science and Technology
Locations (1):
- ROLA, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No